CLINICAL TRIAL: NCT02042768
Title: An Investigation of the Effects of Different Dialysis Prescriptions on Systemic Glucose Metabolism and Mortality in Non-diabetic Peritoneal Dialysis Patients
Brief Title: Observational Study of Glucose Metabolism and How Dialysate Glucose Affects This
Acronym: PD-CRAFT
Status: Completed | Type: Observational
Sponsor: Keele University (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Baxter Healthcare Corporation (Industry); Kidney Cancer UK (Other)
Responsible Party: Sponsor
Other Study IDs: RG-0077-16, 010/12
Record Dates: First submitted 2014-01-10; First posted 2014-01-23 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Glucose Metabolism Disorders
Keywords: Glucose; Dialysate; Peritoneal Dialysis; patients; non-diabetic
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood stored in EDTA for assays including DNA on all PD-CRAFT patients. 10mls blood in EDTA taken during PET on all patients eligible for glucose study.
  30mls of spent dialysate stored in both filtered and unfiltered aliquots on all patients on PD for more than 3 years.
Oversight: Data Monitoring Committee: No

SUMMARY:
Peritoneal Dialysis (PD) is a commonly used treatment for end stage renal failure, and the most commonly used dialysate contains unphysiological amounts of glucose, a high proportion of which is absorbed. Recent analysis of the Global Fluid Study, has established that in non-diabetic prevalent patients on PD a random glucose level is dependent on dialysate glucose load and is a predictor of death. By utilising clinical data and additional biosamples collected for the NIHR funded PD-CRAFT study, the investigators aim to confirm this finding, define the relationship between dialysate glucose exposure according to prescription regimes and glycaemia, define the most useful biomarker to monitor glycaemia , and establish the role that impaired insulin sensitivity plays in blood glucose levels. Furthermore the investigators will explore the hypothesis that insulin resistance is associated with disturbance of the carnitine/acetyl-carnitine equilibrium that might benefit from intra-peritoneal carnitine supplementation.

PD-CRAFT is an observational cohort study of 3000 prevalent PD patients collecting detailed clinical data, including glucose exposure and samples of dialysate. and blood which will be stored in the UK BioCentre. Follow up is for up to 2 years or endpoint (death, technique failure).

Multivariate regression will be used to establish determinants of the non-fasting blood glucose and other measures of glycaemia, in particular different dialysis regimes, (e.g. modality, dwell lengths, fill volumes, and dialysate type and concentration specifically seeking to identify prescriptions that minimise the systemic effects) combined with measures of insulin resistance. The investigators will establish whether blood glucose predicts survival in an adjusted analysis (~300 endpoints needed) using Cox regression and explore the relationship of other biomarkers to survival.

ELIGIBILITY:
Inclusion Criteria:

* On peritoneal dialysis

Exclusion Criteria:

* Not providing informed consent.
* Diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All incident and prevalent non-diabetic peritoneal dialysis patients at centres participating in PD-CRAFT in the UK. PD-CRAFT is designed to oversample patients on PD for longer periods of time.
Sampling Method: Non-Probability Sample
Enrollment: 1451 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Patients will be followed up for the duration of the study period, an expected average of 24 months
  From study entry to date of death from any cause, assessed up to June 2015

SECONDARY OUTCOMES:
Cardiovascular mortality | Patients will be followed up for the duration of the study period, an expected average of 24 months
  From study entry up to date of death from cardiovascular cause, assessed up to June 2015

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lambie, MD, Principal Investigator — Keele University
Locations (1):
- University Hospital of North Staffordshire, Stoke-on-Trent, North Staffordshire, United Kingdom

REFERENCES:
- See also: Study website — http://www.keele.ac.uk/pd-craft/